CLINICAL TRIAL: NCT03813823
Title: Biobehavioral Correlates of Acute Phobic Fear: Proinflammatory, Autonomic, and Neurocognitive Outcomes
Brief Title: Biobehavioral Correlates of Acute Phobic Fear
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Colorado, Boulder (Other)
Responsible Party: Principal Investigator, Alex Kirk, Graduate Student, University of Colorado, Boulder
Other Study IDs: 18-0284
Record Dates: First submitted 2018-12-17; First posted 2019-01-23 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Phobia
MeSH Terms: conditions — Phobic Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood plasma; saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Phobic: Adults aged 18-40 exhibiting high levels of self-reported phobic symptoms to spiders
  Interventions: Behavioral: Fear tasks
- Nonphobic: Adults aged 18-40 exhibiting low levels of self-reported phobic symptoms to spiders
  Interventions: Behavioral: Fear tasks

INTERVENTIONS:
Behavioral: Fear tasks — All participants will be exposed to 5 fear tasks involving spiders, with increasing fear intensity.

SUMMARY:
This study seeks to measure the time course of circulating proinflammatory markers (interleukin-1 beta [IL-1β], interleukin-6 [IL-6], tumor necrosis factor alpha [TNF-α], and C-reactive protein [CRP]) and salivary alpha amylase (sAA) following laboratory fear arousal. Further, this study seeks to implement neurocognitive, physiological, and self-report measures to explore the role of threat sensitivity as a predictor of this response. The broad research question seeks to better understand the relationship between neurocognitive fear and subsequent stress responding elicited by both the immune system (i.e., proinflammatory markers) and autonomic nervous system (i.e., sAA). In light of these aims, the primary outcomes of the current study are the proinflammatory markers (IL-1β, IL-6, TNF-α, CRP), while secondary outcomes consist of sAA, neurocognitive measures (i.e., dot-probe task), physiological correlates (i.e., heart rate, galvanic skin response), and self-report measures.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 40 years old
* Phobic or nonphobic fear of spiders.
* Willing to proceed through 5-stimulus fear hierarchy or maintain 7 or higher subjective units of distress through fear task (see Procedures section).

Exclusion Criteria:

* Lifetime history of serious mental illness
* Lifetime history of intellectual or developmental delays
* Lifetime history of chronic physical or medical illness including blood clotting disorders
* Lifetime history of allergies to latex
* Lifetime history of hormonal replacement therapy
* Lifetime history of blindness
* Lifetime history of blood/injection phobia or aversion to needles/injection (based on IPS-Anx and MQ)
* Substance abuse in the past 2 years
* Cigarette/tobacco use in the past 2 years
* Major depression within the past 12 months
* Traumatic stress within the past 12 months
* Pregnancy within the past 12 months
* Anesthesia within the past 3 months
* Night shift work within the past month
* Use of medication within the past month (except for oral contraception)
* Acute illness or infection within the past month
* Average sleep outside of 6 - 10 hours per night within the past month
* Average intake of 4 or more alcoholic beverages per week
* Average intake of 6 or more cups caffeine per day
* Use of marijuana within the week before the laboratory session
* Use of alcohol within the week before the laboratory session
* Body mass index outside of 18.5 - 24.9 range

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy participants exhibit high or low fear towards spiders.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2019-02-04 (Estimated); Primary Completion 2019-08-01 (Estimated); Study Completion 2019-08-01 (Estimated)

PRIMARY OUTCOMES:
Blood plasma concentration of IL-1 beta | 4 hours
  interleukin-1 beta (pg/mL) via blood draw
Blood plasma concentration of IL-6 | 4 hours
  interleukin-6 (pg/mL) via blood draw
Blood plasma concentration of TNF-alpha | 4 hours
  Tumor necrosis factor-alpha (pg/mL) via blood draw
Blood plasma concentration of CRP | 4 hours
  C-reactive protein (mg/L) via blood draw

SECONDARY OUTCOMES:
Autonomic marker: alpha amylase | 50 minutes
  salivary alpha amylase
Autonomic marker: galvanic skin response | 4 hours
  galvanic skin response (GSR) via Empatica E4 wristband
Autonomic marker: heart rate | 4 hours
  heart rate variability (HRV) via Empatica E4 wristband
Threat sensitivity: neurocognitive task | 10 minutes
  exogenous cueing task via PsychoPy
Threat sensitivity: self-report | 10 minutes
  Clinician-Administered PTSD Scale for DSM-5 (CAPS-5); 6 items (B4, B5, D4, D5, C1, C2) reworded for spider phobia

CONTACTS AND LOCATIONS:
Overall Officials: Alex Kirk, M.A., Principal Investigator — University of Colorado, Boulder; Joanna Arch, Ph.D., Principal Investigator — University of Colorado, Boulder

IPD SHARING:
Plan to Share IPD: Undecided